CLINICAL TRIAL: NCT04974333
Title: Development of an Information Board and Mobile Application for the Care of Type 2 Diabetes at the First Level of Medical Care for the Health Sector in Mexico
Brief Title: Development of an Information Board and Mobile Application for the Care of Type 2 Diabetes
Acronym: SANENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Health Council, Mexico (Other Government)
Collaborators: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-001-20181109
Record Dates: First submitted 2021-06-30; First posted 2021-07-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes type 2; mobile health technology; diabetes control; intervention; lifestyle habits
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile health application (Experimental): Participants assigned to the intervention group will use a mobile application on their smart phones that will assist the patients with their diabetes control, provide and update information on their clinical history, offer a monitoring their nutritional and physical activity habits as well as anthropometric measurements, provide recommendations how to improve on nutritional habits and physical activity behavior, assist in planning and reminding on clinical appointments.
  The duration of the intervention will be 12 months. Each patient will be invited to follow-up visits and measurements each three months (month 3, month 6, month 9 and month 12).
  Interventions: Device: Mobile health application on phone
- Standard care (No Intervention): Participants assigned to the control arm will continue their regular standard diabetes care without mobile health technology assistance.

INTERVENTIONS:
Device: Mobile health application on phone — Patients will use a mobile app on their smart phones
  Arms: Mobile health application

SUMMARY:
The SANENT trial is a primary care-based, prospective, two-arm, randomized controlled, open-label, blinded-endpoint study with the aim to compare a diabetes management strategy using an information board and a mobile application versus standard care in patients with uncontrolled type 2 diabetes. This trial aims to recruit 1440 type 2 diabetes patients during a period of six months until the requested number of participants have been achieved. The total length of the intervention will be one year. The SANENT trial protocol is presented according to Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) recommendations

DETAILED DESCRIPTION:
Trial setting

This trial will be conducted within primary health care practices in three states (Colima, Tlaxcala y Guanajuato) of Mexico. These states were selected because they have a high prevalence of diabetes and have implemented an Electronic Health Record System.

Patient and Public involvement

During the planning phase of the study, a pilot project was carried out evaluating the design and applicability of the information board and mobile application in 31 type 2 diabetes patients. The final intervention was then modified according to the qualitative data received from the patients. the investigators also involved primary healthcare clinicians in the development and evaluation of the information. The results of the study will be made available to all trial participants and participating general practices. Finally, the General Health Council of Mexico who manages the countries public health system is included as collaboration partner in this trial and has been involved in all phases of the design of this study.

Sample size calculations

Considering a difference in HbA1C of 0.5% between the intervention and the control group, a standard deviation of 1.5%, a power of 90% and an alpha of 0.05 (two-sided tests) with a drop-out rate of 25% during the study, a minimum of 504 will be needed in total in each of the three states. Thus, the total number of patients will be 1512.

Screening and recruitment

The participating healthcare centers were selected because they have the most recent version of the Electronic Health Record System that allows linking clinical information to the mobile app and the information board used in this study. In addition, these centers count with the necessary health information system infrastructure. Finally, each of these centers take care of the clinical control of diabetes patients. The primary healthcare workers of the participating centers will screen their type 2 diabetes patient lists and will invite eligible patients. Patients will receive an invitation letter and a leaflet with general information about the study. Eligible patients may also be contacted by phone, emails, or text by the healthcare professionals. Patients will be enrolled for screening and random allocation over a six-month period. During the first visit of the screening phase, the eligibility criteria and medical record will be revised by the healthcare professionals. In case the patient is potentially eligible, the patient will be invited to the study upon obtaining informed consent. Before the next screening visit, the HbA1C of the patient will be measured to complete the eligibility assessment. Once the diagnosis of uncontrolled type 2 diabetes has been made, all other baseline measurements and laboratory tests will be conducted.

Random allocation

This trial will use a parallel group design, randomizing patients to either the intervention or the control arm by a computer-generated sequence with an allocation ratio of 1:1. The randomization of the study participants will be done after having provided consent and when all baseline assessments have been completed to minimize reporting and selection bias.

Random allocation will be done using a validated secure web-based randomization operated by a data manager, not involved in the patient recruitment, located at the Autonomic University of Mexico. This will ensure concealment of the treatment sequence up to the allocation. The treatment sequence will be generated by a computer-generated sequence of random numbers. Allocation will be carried out with an algorithm to ensure groups are balanced for important baseline prognostic and other factors: study site, age (<65/≥65 years), sex (male/female), duration of diabetes (<5 years/≥5 years) and number of medications (<5/≥5) which are considered as a key prognostic variable for the primary outcome of this trial. The treatment allocation codes will be concealed in sequentially numbered envelopes that will be opened each time a patient will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Men and women treated for type 2 diabetes with an HbA1C>8.5%;
* ≥20 years-of-age;
* Signed up for diabetes treatment and control in one of the participating primary healthcare practices.
* Having access to a mobile phone (or having a family member who will help them in sending, understanding, and retrieving messages and information provided in Spanish language through the mobile application)

Exclusion Criteria:

* Participants who are pregnant, within 3 months postpartum or planning pregnancy during the trial;
* Breastfeeding;
* Serious medical condition (i.e. dialysis treatment);
* Having been admitted to hospital within the last 3 months for hyperglycemia or hypoglycemia;
* Not permanent residents of the states where the study is conducted.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1512 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 12 months
  Change in HbA1C

SECONDARY OUTCOMES:
Blood lipids changes | 12 months
  Changes in serum cholesterol, LDL, HDL cholesterol, triglycerides
Blood pressure changes | 12 months
  Changes in systolic and diastolic blood pressure
Body mass index | 12 months
  Changes in body mass index (kg/m2)
Treatment compliance change | 12 months
  Treatment compliance using Morisky scale. The Morisky scale is a validated scale designed to estimate the risk of medication non-adherence. The scale consists of eight questions, first seven items having a dichotomous answer (yes/no) that indicates adherent or non-adherent behaviour. For item 8, a patient can choose an answer on a 5-point Likert scale, expressing how often happens that a patient does not take his medications. The Morisky scores can range from 0 to 8 points.
Mental health improvement | 12 months
  Depression will be measured using the Beck questionnaire. The Beck questionnaire adda up the score reported for each of the 21 questions ranging from zero to three. Each answer is scored on a scale value of 0-3. Measures of 0-9 indicates that a person is not depressed, 10-18 indicates mild-moderate depression, 19-29 indicates moderate-severe depression and 30-63 indicates severe depression.
Physical activity changes | 12 months
  Changes in physical activity will be assessed using the International Physical Activity Questionnaire. The International Physical Activity Questionnaire allows to estimate the overall total physical activity metabolic equivalents-minutes/week score. All activities are converted into minutes before calculating metabolic equivalent minutes. To calculate metabolic equivalents minutes a week the metabolic equivalents value given is multiplied (remember walking = 3.3, moderate activity = 4, vigorous activity = 8) by the minutes the activity was carried out and again by the number of days that that activity was undertaken. The higher the metabolic equivalent-minutes/week score, the more activity the participant is.
Changes in albumin to creatine ratio | 12 months
  Changes in kidney function will be measured using the albumin to creatine ratio. A ratio of albumin (mcg/L) to creatinine (mg/L) of less than 30 is normal; a ratio of 30-300 signifies microalbuminuria and values above 300 are considered as macroalbuminuria.
Quality of life changes | 12 months
  Short Form 36 questionnaire assessing changes in quality of life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Waist circumference | 12 months
  Change in waist circumference (measured in cm)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Cisneros Gonzalez, MD, Principal Investigator — Consejo General de Salud
Locations (3):
- Mexico (3):
  - Coordinacion Clinica de Educacion e Investigacion en Salud Medicina Familiar, Mexico City, Mexico City
  - Unidad de Medicina Familiar 33, Chihuahua City
  - Establecimiento salud: Centro de Salud Urbano Zona Oriente "La Vurgencita", Colima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barengo NC, Apolinar LM, Estrada Cruz NA, Fernandez Garate JE, Correa Gonzalez RA, Diaz Valencia PA, Gonzalez CAC, Rodriguez JAG, Gonzalez NC; SANENT Study Group. Development of an information system and mobile application for the care of type 2 diabetes patients at the primary care level for the health sector in Mexico: study protocol for a randomized controlled, open-label trial. Trials. 2022 Apr 4;23(1):253. doi: 10.1186/s13063-022-06177-0. PMID 35379298